CLINICAL TRIAL: NCT01878318
Title: Open Label Study to Describe the Effect of Tocilizumab in Combination With MTX in the Evolution of Articular Damage (Synovitis/Osteitis and Erosions) Evaluated by MRI in the Hand of Patients With Moderate to Severe Rheumatoid Arthritis (RA) and Inadequate Response to Non-biological DMARDs
Brief Title: A Study of The Effect of RoActemra/Actemra (Tocilizumab) in Combination With Methotrexate on Articular Damage in The Hand in Patients With Moderate to Severe Rheumatoid Arthritis Who Have an Inadequate Response to Non-Biological DMARDs
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28204
Record Dates: First submitted 2013-06-06; First posted 2013-06-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; tocilizumab

ARMS (1):
- RoActemra/Actemra (Experimental)
  Interventions: Drug: methotrexate; Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: methotrexate — stable dose
Drug: tocilizumab [RoActemra/Actemra] — 8 mg/kg intravenously every 4 weeks, 24 weeks

SUMMARY:
This open-label, single arm study will evaluate the effect of RoActemra/Actemra in combination with methotrexate on articular damage in the hand (synovitis/osteitis and erosions) in patients with moderate to severe rheumatoid arthritis who have an inadequate response to non-biological disease-modifying ante-rheumatic drugs (DMARDs). Patients will receive RoActemra/Actemra 8 mg/kg intravenously every 4 weeks for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Diagnosis of rheumatoid arthritis according to ACR/EULAR classification (2010) of >/= 6 months duration
* Active moderate to severe rheumatoid arthritis (DAS >/= 3.2)
* Swollen joint count (SJC) >/= 6, tender joint count >/= 8
* Synovitis in the dominant hand
* Inadequate response to stable dose of a non-biological DMARD for at least 3 months
* Oral corticosteroids must have been on stable dose for at least 25 out of 28 days before first dose of study drug
* Patient on outpatient treatment

Exclusion Criteria:

* Major surgery (including joint surgery) in the 8 weeks prior to screening, or planned major surgery within 6 months of randomization
* Rheumatic autoimmune disease other than rheumatoid arthritis
* American College of Rheumatology (ACR) functional class IV
* History of or current inflammatory joint disease other than rheumatoid arthritis
* Previous inadequate response to a biologic DMARD; prior biologic therapy for no longer than 1 month is allowed if discontinued for reasons of tolerability at least 6 months prior to study recruitment
* Intra-articular or parenteral corticosteroids within 6 weeks prior to study start
* Inadequate hematologic, renal or liver function
* Positive for hepatitis B, hepatitis C or HIV infection
* Pregnant or lactating women
* History of severe allergic reactions or anaphylaxis to human, humanized or mural monoclonal antibodies
* Current infections or history of recurrent infections
* History of or currently active primary or acquired immunodeficiency
* Active tuberculosis requiring treatment in the previous 3 years
* Body weight > 150 kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Change in extent and degree of synovitis in the hand assessed by MRI according to the OMERACT RAMRIS scale | from baseline to Week 24

SECONDARY OUTCOMES:
Radiological changes in the hand according to the modified Sharp scale | from baseline to Week 24
Change in Ritchie articular index | from baseline to Week 24
Proportion of patients with American College of Rheumatology (ACR 20/50/70) response at Weeks 12 and 24 | Weeks 12 and 24
Change in pain: Visual analogue scale (VAS) | from baseline to Week 24
Change in disability: Stanford Health Assessment Questionnaire | from baseline to Week 24
Change in FACIT-fatigue questionnaire | from baseline to Week 24
Change in disease activity: Disease activity score 28 - erythrocyte sedimentation rate (DAS28-ESR) | from baseline to Week 28
Change in C-reactive protein | from baseline to Week 24
Change in immunologic parameters: Rheumatic factor/anti-CCP | from baseline to Week 24
Safety: Incidence of adverse events | approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche